CLINICAL TRIAL: NCT01285115
Title: Phase 3 The Comparative Clinical Study of Gamisoyosan on Anxiety of Generalized Anxiety Disorder According to Dosage Form : A Randomized, Double Blind, Parallel-controlled Trial
Brief Title: The Comparative Clinical Study of Gamisoyosan on Anxiety of Generalized Anxiety Disorder According to Dosage Form
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: the president of Korea Health Industry Development Institute, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B082005
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2010-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized anxiety disorder; Jingji-zhengchong; Gamisoyosan; anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo; corn flour, (Placebo Comparator): * raw material total contents(500㎎) cornstarch 50.0%(250.0㎎), 당수화물 49.45%(247.25㎎), caramel pigment 0.5%(2.5㎎), SsangHwa fragrance 0.05%(0.25㎎)
  * shape, type: extract(brown)
  * usage, content: adults;three times a day each sack taken before or between meals
  * dose, standard: for each sack 7.67g
  * storage : airtight container, stored in room temperature
  * expiration date : after manufacture 36 month
  * macufacturing company: KyungBangnShinYak inc.
  Interventions: Drug: Placebo
- Gamisoyosan extract (Active Comparator): * name of product: KyungBangn-Gamisoyosan-x-gwarip
  * standard code for item : 200005799
  * shape, type: extract(grayish brown)
  * usage, content : adults;three times a day , each sack taken before or between meals
  * dose, standard: 7.67g for each sack
  * storage : airtight container, stored in room temperature expiration date : after manufacture 36 month macufacturing company: KyungBangnShinYak inc.
  Interventions: Drug: KyungBangn-Gamisoyosan-x-gwarip
- Gamisoyosan extract powder (Active Comparator): * name of product: KyungBangn Gamisoyosan
  * standard code for item: 200005591
  * shape, type: powder(brown)
  * usage, content: adults;three times a day each sack taken before or between meals
  * dose, standard: 7.67g for each sack
  * storage : airtight container, stored in room temperature
  * expiration date : after manufacture 36 month
  * macufacturing company: KyungBangnShinYak inc.
  Interventions: Drug: KyungBangn Gamisoyosan

INTERVENTIONS:
Drug: Placebo — AC 30 min, three times a day each sack taken before or between meals, 7.67g for each sack, 8 weeks.
  Arms: Placebo; corn flour,
Drug: KyungBangn-Gamisoyosan-x-gwarip — AC 30 min, three times a day each sack taken before or between meals, 7.67g for each sack, 8 weeks.
  Other Names: standard code for item : 200005799
  Arms: Gamisoyosan extract
Drug: KyungBangn Gamisoyosan — AC 30 min, three times a day each sack taken before or between meals, 7.67g for each sack, 8 weeks.
  Other Names: standard code for item: 200005591
  Arms: Gamisoyosan extract powder

SUMMARY:
In this randomized, double blinded, Parallel-controlled study, the investigators planned to give Gamisoyosan extract, Gamisoyosan extract powder or controlled medication on Anxiety of generalized anxiety disorder according to dosage form.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20-65
* (Structured Clinical Interview for DSM-Ⅳ Axis Ⅰ Disorder, SCID-Ⅰ) subjects who meet Structured Clinical Interview for DSM-Ⅳ Axis Ⅰ Disorder, SCID-Ⅰof generalized anxiety disorder

Exclusion Criteria:

* Currrent or past history of delusions, halucination
* Past history of at least one manic episode, hypomanic episode, or mixed episode
* Current or past history of alcohol abuse or alcohol dependence history
* Taking substances(e.g. antianxiety drugs, antidepressant, antipsychotic drug, steroids, female hormonal drug, L-dopa, digitalis, bromide, cyclosporin, disulfiram, isoniazid, yohimbine) which might affect symptoms
* Medical conditions(e.g. myocardial infarction,brain tumor, multiple sclerosis, pancreatic disease, hyperthyroidism, hypothyroidism, Addison disease, Cushing disease, rheumarthritis, cancer, CVA, epilepsy, anemia, pituitarium disease, Vit B12 deficiency disease, PMS) that might affect symptoms
* Current with hepatoma, hepatic cirrhosis, chronic renal failure, congestive heart failure
* Pregnancy, lactation, women not using medically accepted means of birth control
* Considered not apt to carry out clinical trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2008-12; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale(HAM-A) | 8 weeks
  The HAM-A (Hamilton Anxiety Scale) is a widely used interview scale that measures the severity of a patient's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory(STAI) | 8 weeks
  The State-Trait Anxiety Inventory (STAI) was initially conceptualized as a research instrument for the study of anxiety in adults. It is a self-report assessment device which includes separate measures of state and trait anxiety.
Beck Depression Inventory(BDI) | 8 weeks
  BDI is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. Each question has a set of at least four possible answer choices, ranging in intensity. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity.
Symptom Checklist-90-Revised(SCL-90R) | 8 weeks
  The Symptom Checklist-90-R (SCL-90-R) is a relatively brief self-report psychometric instrument (questionnaire). It is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It is also used in measuring the progress and outcome of psychiatric and psychological treatments or for research purposes.
WHO Quality of Life Abbreviated(WHOQOL-BREF) | 8 weeks
  Quality of life is used to evaluate the general well-being of individuals and societies.
Heart Rate Variability(HRV) | 8 weeks
  Heart rate variability (HRV) is a physiological phenomenon where the time interval between heart beats varies. It is measured by the variation in the beat-to-beat interval.
PSWQ | 8 weeks
  The Penn State Worry Questionaire is a 16-item inventory assess worry and anxiety
GSES | 8 weeks
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
RSE | 8 weeks
  Rosenberg Self-Esteem Scale is questionnaire that popular lore recognizes just "high" self-esteem and "low" self-esteem, the Rosenberg Self-Esteem Scale quantify it in more detail, and feature among the most widely used systems for measuring self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: In-Chul Jung, Ph.D, Principal Investigator — Oriental Hospital of Daejon University
Locations (1):
- Oriental Hospital of Daejon University, Daejeon, Choong-Chung-Do, South Korea